CLINICAL TRIAL: NCT02890472
Title: Research of Thymix Dysgenesis in Prenatal Examination of Deletion 22q11 Syndrome
Brief Title: Prenatal Examination of Deletion 22q11 Syndrome : Thymic Dysgenesis THYMI Study
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/EM-01
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: 22q11 Deletion Syndrome Di George Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- prenatal diagnosis of a fetal 22q11 deletion syndrome

SUMMARY:
22q11.2 microdeletion seems the prenatally under-diagnosed . Indeed , there is a mismatch between the series on the heart rate of 22q11.2 antenatal 84% against 30% in the adult series despite a perinatal mortality of 16% suggesting opportunities for improvement in the prenatal diagnosis of fetus with a microdeletion 22q11.2 , especially without heart disease

ELIGIBILITY:
Inclusion Criteria:

* all prenatal diagnosis with FISH or CGH array of a fetal 22q11 deletion syndrome during the inclusion period.
* The pregnancy follow-up should be done one of the 44 french fetal medicine unit.
* Sonographic picture of 3 vessels slides should be communicated for independent review.

Exclusion Criteria:

* no sonographic picture available

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prenatal diagnosis of a fetal 22q11 deletion syndrome
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Thymic thoracic ratio " measurement on sonographic picture of the fetal 3 vessels slides will be done by independent investigator. | day 0

CONTACTS AND LOCATIONS:
Locations (1):
- CHUNimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: Yes